CLINICAL TRIAL: NCT03428906
Title: Effects of Intranasal Oxytocin on Male's Functional Brain Network in Resting-state and Tasks
Brief Title: Effects of Intranasal Oxytocin on Functional Brain Network in Resting-state and Tasks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Normal University (Other)
Responsible Party: Principal Investigator, ma, yina, Principal Investigator, Beijing Normal University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IN-OT functional network
Record Dates: First submitted 2018-02-04; First posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Healthy
Keywords: intranasal oxytocin; functional brain network; multiple tasks; resting state
MeSH Terms: interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The study utilized a randomized, double-blind, PBO controlled, within-subject design, in which each participant was tested under two acute treatment conditions separated by at least 1 wk wash-out period.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxytocin (Experimental): Oxytocin (OXT), a neuropeptide produced in the hypothalamus, is a key modulator of complex socioaffective responses including affiliation, social approach and attachment, stress and anxiety. Subjects receiving an intranasal spray of OXT (8 IU or 13.44 mg; Syntocinon-spray; Novartis, Switzerland) .
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Placebo contains all ingredients except for the peptide in three puffs of 1.33 IU per 2.24mg nostril.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — intranasally administrated
  Arms: Oxytocin
Drug: Placebo — intranasally administrated
  Other Names: Saline
  Arms: Placebo

SUMMARY:
To investigate whether and how intranasal oxytocin of 8IU treatment will alter the topology of functional brain network in resting-state and multiple tasks in healthy males.

DETAILED DESCRIPTION:
In a randomized, double-blind, cross-over, placebo controlled design, healthy male volunteers receive intranasal oxytocin or placebo prior to functional magnetic resonance imaging.Subjects will then go through a decision making task, a emotion judgement task and an eight-minute resting-state scan in MRI scanner to investigate whether and how intranasal oxytocin alter the topology of functional brain network in resting-state and multiple tasks in healthy males. State anxiety and mood are measured before and after experiment as covariates to be controlled.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects without past or current psychiatric or neurological disorders

Exclusion Criteria:

* with MRI Contraindications

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — we opted to recruit only males for the present study.
Enrollment: 34 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2017-09-12 (Actual)

PRIMARY OUTCOMES:
Functional network organization alterations in brain under resting state fMRI after drug administration | 70~85 minutes after drug administration
  Using seed-based and network level functional connectivity analysis, as well as graph theory analysis , functional network organization in brain under eight minutes resting state will be detected and compared between oxytocin and placebo group.
Behavior,brain activities and representation patterns in the emotional judgement task after drug administration | 60~75 minutes after drug administration
  Friend or Foe Task is used to measure the verbal versus nonverbal emotional judgement of subjects. Both the response of subjects and the brain activity are recorded in the task. How oxytocin influences the relationship between subjects' behavior and representation pattern of emotional judgement will be investigated through RSA(representation similarity analysis) of brain pattern.
Behavior, dynamics brain activities and networks in the model-based decision making task after drug administration | 35~60 minutes after drug administration
  Two-Stage Decision Making Task is used to measure the model-based and model-free decision making process of subjects. The degree of model-based will be calculated by Computational modelling of Subjects' decision making process, and entering as modulation parameter in the OT effect on dynamic brain seed-based and network-based connectivity pattern.
Relationship of functional network organization in brain across resting state and task-based fMRI after drug administration | 60~85 minutes after drug administration
  The functional brain activity in resting state, emotional judgement and decision making task will be compared. Both the functional segregation and integration will be measured using graph theory and network connectivity analysis to discover the OT effect on brain network organization across multiple cognitive states.

CONTACTS AND LOCATIONS:
Overall Officials: Yina Ma, PhD, Principal Investigator — School of Brain and Cognitive Sciences, Beijing Nornal University
Locations (1):
- School of Brain and Cognitive Sciences, Beijing Nornal University, Beijing, Beijing Municipality, China